CLINICAL TRIAL: NCT04952558
Title: Diagnostic Lag Time Among Egyptian Inflammatory Bowel Diseased Patients
Brief Title: Delayed Diagnostic Time& Inflammatory Bowel Diseased Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Bahaa osman taha, assistant lecturer, Assiut University
Other Study IDs: ESIBD1989BAHAA
Record Dates: First submitted 2021-06-28; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Lag time; inflammatory bowel disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cross sectional observational study: Cross sectional observational study will be conducted among 700 patients of Egyptian inflammatory bowel diseased patients for different regions
  Detailed history will be taken from all included patients focus on
  * age ,sex , special habit ,residence .
  * education level -socioeconomic status
  * type of the inflammatory bowel disease
  * lag time for reaching the proper diagnosis of inflammatory bowel disease which definite as time from the first symptoms presentation to reaching definite diagnosis
  * symptoms that causing patients seeking medical advice
  * number of Inflammatory bowel diseased patients referred for first time from surgeons
  * number of patients have perianal symptoms
  * number of patients have previous history of appendicectomy

SUMMARY:
Introduction The incidence of inflammatory bowel disease [IBD] is increasing worldwide. Both Crohn's disease [CD] and ulcerative colitis [UC] are therefore becoming an important public health issue[1] The IBD is characterized by chronic intestinal inflammation, which can cause bowel damage and intestinal complications primarily depending on the duration and severity of the inflammation[2] The diagnosis of inflammatory bowel diseases (IBD) is often established following considerable delay due to nonspecific and inconsistent symptoms. In previous western studies, the delayed diagnosis was associated with poor outcome in patients with Crohn's disease (CD).[2] Timely diagnosis is not only important for the patients themselves but has also become a relevant public health issue due to the rising incidence of IBD worldwide[3] Patients and methods Cross sectional observational study will be conducted among 700 patients of Egyptian inflammatory bowel diseased patients for different regions Aim of the study

1. Estimate time delay for diagnosis of Egyptian inflammatory bowel diseased patients
2. compare the delay time for diagnosis of Egyptian inflammatory bowel diseased patients globally

DETAILED DESCRIPTION:
diagnostic Lag time among Egyptian inflammatory bowel diseased patients

Introduction The incidence of inflammatory bowel disease [IBD] is increasing worldwide. Both Crohn's disease [CD] and ulcerative colitis [UC] are therefore becoming an important public health issue[1] The IBD is characterized by chronic intestinal inflammation, which can cause bowel damage and intestinal complications primarily depending on the duration and severity of the inflammation[2] The diagnosis of inflammatory bowel diseases (IBD) is often established following considerable delay due to nonspecific and inconsistent symptoms. In previous western studies, the delayed diagnosis was associated with poor outcome in patients with Crohn's disease (CD).[2] Timely diagnosis is not only important for the patients themselves but has also become a relevant public health issue due to the rising incidence of IBD worldwide[3] Abdominal pain is the most prevalent initial chief complaint in patients with CD; however, it is also a common symptom of other digestive disorders, such as irritable bowel syndrome may the pain is not severe, it is easily regarded as trivial, and the diagnosis may be missed because the tests needed for the diagnosis of IBD are not performed. [4] A delayed diagnosis of CD may incur high medical cost in patients who develop aggressive disease that requires treatment with anti-TNFα agents[5] Aim of the study

1. Estimate time delay for diagnosis of Egyptian inflammatory bowel diseased patients
2. compare the delay time for diagnosis of Egyptian inflammatory bowel diseased patients globally
3. studing risk factors that causing diagnostic delay among Egyptian inflammatory bowel diseased patients the time
4. frequency of diagnosed complicated inflammatory bowel diseased as first time presentation

Patients and methods Cross sectional observational study will be conducted among 700 patients of Egyptian inflammatory bowel diseased patients for different regions

Inclusion criteria Egyptian inflammatory bowel diseased patients above the age of 18 years with definite diagnosis based on clinical ,endoscopic ,histological basis

Detailed history will be taken from all included patients focus on

* age ,sex , special habit ,residence .
* education level -socioeconomic status
* type of the inflammatory bowel disease
* lag time for reaching the proper diagnosis of inflammatory bowel disease which definite as time from the first symptoms presentation to reaching definite diagnosis
* symptoms that causing patients seeking medical advice
* number of Inflammatory bowel diseased patients referred for first time from surgeons
* number of patients have perianal symptoms
* number of patients have previous history of appendicectomy
* physicians numbers that visited by the patients to reaching the diagnosis
* ileal intubation at first time colonoscopy
* number of patients change their diagnosis from ulcerative colitis to Crohn's disease
* type of radiological assessment of the examined patients

Exclusion criteria Inflammatory bowel diseased Patients below 18 years old

Ethical consideration:

consent will be taken from all participating patients and must be approved by the ethical committee

References :

1. E. V. Loftus, "Clinical epidemiology of inflammatory bowel disease: Incidence, prevalence, and environmental influences," Gastroenterology, vol. 126, no. 6, pp. 1504-1517, 2004, doi: 10.1053/j.gastro.2004.01.063.
2. D. W. Lee et al., "Diagnostic delay in inflammatory bowel disease increases the risk of intestinal surgery," World J. Gastroenterol., vol. 23, no. 35, pp. 6474-6481, Sep. 2017, doi: 10.3748/wjg.v23.i35.6474.
3. S. R. Vavricka et al., "Systematic evaluation of risk factors for diagnostic delay in inflammatory bowel disease," Inflamm. Bowel Dis., vol. 18, no. 3, pp. 496-505, Mar. 2012, doi: 10.1002/ibd.21719.
4. G. Novacek et al., "Diagnostic delay in patients with inflammatory bowel disease in Austria," Wien. Klin. Wochenschr., vol. 131, no. 5-6, pp. 104-112, Mar. 2019, doi: 10.1007/s00508-019-1451-3.
5. L. Cantoro et al., "The Time Course of Diagnostic Delay in Inflammatory Bowel Disease Over the Last Sixty Years: An Italian Multicentre Study," J. Crohn's Colitis, vol. 11, no. 8, pp. 975-980, Aug. 2017, doi: 10.1093/ecco-jcc/jjx041.

ELIGIBILITY:
Inclusion Criteria:

Egyptian inflammatory bowel diseased patients above the age of 18 years with definite diagnosis based on clinical ,endoscopic ,histological basis

-

Exclusion Criteria:

Inflammatory bowel diseased Patients below 18 years old

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cross sectional observational study will be conducted among 700 patients of Egyptian inflammatory bowel diseased patients for different regions
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
measure time delay for diagnosis of Egyptian inflammatory bowel diseased patients | 2 months
  duration in months from the first symptoms appearance till the definite diagnosis
compare the delay time for diagnosis of Egyptian inflammatory bowel diseased patients globally | 4 months
  difference in months between global delay and Egyptian delay for diagnosis of inflammatory bowel disease

CONTACTS AND LOCATIONS:
Locations (1):
- Bahaa Osman Taha, Asyut, Egypt